CLINICAL TRIAL: NCT05102734
Title: Trial of a Topical Nitroglycerin Challenge to Detect Reversible Microcirculatory Dysfunction in Patients With Circulatory Shock.
Brief Title: Physiologic Effect of Topical Nitroglycerin on Microcirculation Capacity in Patients With Circulatory Shock.
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 843615
Record Dates: First submitted 2021-10-21; First posted 2021-11-01 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Circulatory Shock; Cardiovascular Shock
MeSH Terms: conditions — Shock; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Topical nitroglycerin: A topical nitroglycerin solution will be applied to the area of interest
  Interventions: Drug: Nitroglycerin Topical Product

INTERVENTIONS:
Drug: Nitroglycerin Topical Product — Topical nitroglycerin solution

SUMMARY:
This is an open-label, single center, trial that will enroll up to 25 participants with circulatory shock after cardiac surgery. Participants will be administered a topical sublingual nitroglycerin solution and assessed for changes microcirculatory blood flow using incident dark field microscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients receiving elective CABG or valvular surgery requiring cardiopulmonary bypass
* Receiving postoperative catecholamine therapy to maintain a MAP > 65mmHg, cardiac index > 2 despite initial fluid resuscitation
* Invasive hemodynamic monitoring

Exclusion Criteria:

* Surgical hemorrhage
* Unable to tolerate sublingual microcirculatory flow imaging
* Known intolerance or allergy to nitroglycerin
* Inadequate microcirculation imaging (based on Massey Score)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiovascular surgery
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C. Greenwood, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of the Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication of demographics, study drug effects, changes in hemodynamics and microcirculation. Limited, de-identified data can be made available upon request.
Supporting Information: CSR
URL: https://zenodo.org/record/5768720

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment completed between August 1 and October 30, 2021.
Pre-assignment Details: 20 patients were enrolled to obtain preoperative control microcirculation measurements only. 20 additional patients would be needed for the NTG challenge. NTG patients were enrolled prior to surgery, but not included if they did not meet postop inclusion criteria.
Groups:
- Preoperative Control Group: Subjects planned for elective cardiovascular surgery were enrolled to measure baseline microvascular function by sublingual incident darkfield microscopy imaging.
Period: Overall Study
Arm/Group | Topical Nitroglycerin | Preoperative Control Group
Started | 24 | 20
Completed | 20 | 20
Not Completed | 4 | 0
Not completed — Did not require vasopressors | 1 | 0
Not completed — Did not have functioning PA catheter | 1 | 0
Not completed — Inadequate video quality | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Preoperative Control Group: 20 subjects planned for elective cardiovascular surgery were enrolled to measure baseline microvascular function by sublingual incident darkfield microscopy imaging.
- Total: Total of all reporting groups
Arm/Group | Topical Nitroglycerin | Preoperative Control Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (9) | 67 (11) | 65 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 18 | 18 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Perfused Vessel Density (PVD)
Description: Estimate of functional capillary density.
Time Frame: Preoperative Control Group: assessed once preoperatively. For the topical nitroglycerin group, PVD measurements were obtained after surgery (baseline), then 3-minutes and 30-minutes after topical nitroglycerin administration.
Population: Sublingual microcirculation measurements were obtained in a preoperative control group to serve as a "healthy" control measurement to compare against measurements in patients with shock. The preoperative control group only had one PVD measurement taken. Sublingual microcirculation measurements in the topical nitroglycerin group were measured after surgery (baseline), then 3-minutes and 30-minutes after NTG solution application.
Measure: Mean (Standard Deviation); unit: mm/mm^2
Groups:
- Topical Nitroglycerin Group Postop Baseline: Postop baseline measurement of PVD.
  A topical nitroglycerin solution will then be applied to the sublingual space.
- Topical Nitroglycerin Group 3-minutes Post-NTG: PVD response 3 minutes after topical NTG solution application.
- Topical Nitroglycerin Group 30-minutes Post-NTG: PVD measured 30 minutes after topical NTG solution application.
Arm/Group | Preoperative Control Group | Topical Nitroglycerin Group Postop Baseline | Topical Nitroglycerin Group 3-minutes Post-NTG | Topical Nitroglycerin Group 30-minutes Post-NTG
Number analyzed (Participants) | 20 | 20 | 20 | 20
mm/mm^2 | 24.81 (3.51) | 20.44 (3.38) | 26.41 (3.50) | 21.88 (3.84)

2. Secondary Outcome: Mean Arterial Pressure
Description: Mean arterial blood pressure
Time Frame: MAP was recorded for the control group, then for the NTG group at postoperative baseline, 3-minutes and 30-minutes after topical NTG application.
Population: Same groups as the primary outcome.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Topical Nitroglycerin Group 3-minutes Post-NTG: PVD response 3 minutes after NTG solution application.
- Topical Nitroglycerin Group 30-minutes Post-NTG: PVD 30 minutes after NTG solution application.
Arm/Group | Preoperative Control Group | Topical Nitroglycerin Group Postop Baseline | Topical Nitroglycerin Group 3-minutes Post-NTG | Topical Nitroglycerin Group 30-minutes Post-NTG
Number analyzed (Participants) | 20 | 20 | 20 | 20
mmHg | 95.85 (11.67) | 71.05 (5.92) | 70.35 (6.8) | 74.4 (7.19)

3. Secondary Outcome: Cardiac Index
Description: Cardiac output relative to patients body surface area
Time Frame: Cardiac output was measured for the control group, then for the NTG group at postoperative baseline, 3-minuts, and 30-minutes after topical NTG application
Population: Same groups as the primary outcome
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Preoperative Control Group | Topical Nitroglycerin Group Postop Baseline | Topical Nitroglycerin Group 3-minutes Post-NTG | Topical Nitroglycerin Group 30-minutes Post-NTG
Number analyzed (Participants) | 20 | 20 | 20 | 20
L/min/m^2 | 2.54 (0.79) | 2.85 (0.81) | 2.88 (0.9) | 2.83 (0.76)

4. Secondary Outcome: Central Venous Pressure
Description: surrogate measure for right atrial pressure
Time Frame: CVP was recorded for the control group, then for the NTG group at postoperative baseline, 3-minutes, and 30-minutes after topical NTG application
Population: Same as the primary outcome
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Preoperative Control Group | Topical Nitroglycerin Group Postop Baseline | Topical Nitroglycerin Group 3-minutes Post-NTG | Topical Nitroglycerin Group 30-minutes Post-NTG
Number analyzed (Participants) | 20 | 20 | 20 | 20
mmHg | 16.7 (5.24) | 9.35 (3.79) | 9.15 (3.25) | 9.16 (3.11)

ADVERSE EVENTS:
Time Frame: Preoperative Control Group: During pre-operative imaging Topical Nitroglycerin Group: At postoperative baseline imaging through 30-minutes after topical nitroglycerin application
Groups:
- Post-NTG Challenge: PVD response after NTG challenge
Arm/Group | Topical Nitroglycerin | Preoperative Control Group | Post-NTG Challenge
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT05102734/Prot_SAP_000.pdf